CLINICAL TRIAL: NCT06693258
Title: A Comparative Study of Transaxillary Robotic Thyroidectomy Versus Standard Open Thyroidectomy
Brief Title: Study of Transaxillary Robotic Thyroidectomy Versus Standard Open Thyroidectomy: Prospective, Comparative Single-Center Study
Acronym: CARTO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Bizet (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024-A01697-40
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Carpal Tunnel Surgery

STUDY DESIGN:
Intervention Model Description: Prospective, Comparative, Monocentric Study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): thyroidectomy by robotic surgery via axillary approach
  Interventions: Procedure: thyroidectomy by robotic surgery via axillary approach
- Control group (Active Comparator): thyroidectomy by standard conventional surgery
  Interventions: Procedure: thyroidectomy by standard conventional surgery

INTERVENTIONS:
Procedure: thyroidectomy by robotic surgery via axillary approach — thyroidectomy
  Arms: Experimental group
Procedure: thyroidectomy by standard conventional surgery — thyroidectomy by standard conventional surgery
  Arms: Control group

SUMMARY:
The aim of our study is to evaluate the two surgical approaches, standard thyroidectomy and robotic thyroidectomy, in terms of postoperative pain management, scar quality, quality of life, as well as the occurrence of postoperative complications (hypocalcemia, compressive cervical hematoma and nerve stimulation)

ELIGIBILITY:
Inclusion Criteria:

* Subject aged over 20 years
* Referred for a thyroidectomy (total or partial)
* Absence of participation in another clinical study
* Subject affiliated to a social security scheme or beneficiary of such a scheme
* Accepts the completion of the various study questionnaires

Exclusion Criteria:

* Patient under 20 years of age.
* Patients who have undergone combined radical cervical lymph node dissection
* Patient with a postoperative wound problem
* Patient with an underlying systemic disease that may influence the wound healing process
* Unable to undergo medical follow-up for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the post-operative quality of life at D30 between the two groups | day 30
  thyca-Qol

SECONDARY OUTCOMES:
Total dysphagia score between the two groups | Day7, Day30 and 3 months
  EAT-10 scale
Quality of the scar between the two groups | day 30
  Vancouver scale
Assess the functional recovery of the vocal cords | day 7 and day 30
  fibroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- clinique Bizet, Paris, France

IPD SHARING:
Plan to Share IPD: No